CLINICAL TRIAL: NCT03742739
Title: Intraoperative Ventilatory Leak Flow to Predict Prolonged Alveolar Air Leak After Lung Resection Surgery: a Prospective Study
Brief Title: Predictive Value of Intraoperative Ventilatory Leak Flow in Prolonged Alveolar Air Leak After Lung Resection Surgery
Acronym: AIR-LEAK
Status: Completed | Type: Observational
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Other Study IDs: UF 7700
Record Dates: First submitted 2018-11-08; First posted 2018-11-15 (Actual); Last update posted 2021-10-19 (Actual); Status verified 2021-03

CONDITIONS: Pronlongated Alveolar Air Leak (PAAL)

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
After lung resection surgery, patients usually receive a postoperative pleural drain. Prolongated alveolar air leak (PAAL) is a frequent complication after lung surgery (6 to 26% of patients), defined by the European Society of Thoracic Surgeons (ESTS) as a duration of drainage greater than or equal to five days. PAAL is most often due to prolongated bubbling of the drain. Prolonged drainage is a leading cause of prolongated hospital stay, increasing care costs.

The risk of prolongated drainage can not be predicted with sufficient accuracy. Existing risk scores for PAAL do not take into account the intraoperative ventilatory leakage (IVL). IVL is a parameter displayed on the ventilator (anaesthetic machine that make the patient breathing during surgical procedure). There is new evidences suggesting that IVL could predict the risk of PAAL after lung resection surgery, but these data have to be supplemented by a well conducted prospective study.

ELIGIBILITY:
Inclusion criteria:

* To be 18 years old or older
* To be of French nationality or native from an European country affiliated to the French health care system
* To be scheduled for pulmonary resection surgery by videothoracoscopy or thoracotomy in the center of the study

Exclusion criteria:

* Patient minor, or major under legal protection, or enable to give consent
* Refusal or consent withdrawal
* No pulmonary resection or no pleural drain at the end of the surgical procedure (decided by the surgical team)
* Postoperative pleural fistula

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients scheduled for pulmonary resection surgery by videothoracoscopy or thoracotomy (including pulmonary wedge resection, segmentectomy, lobectomy, bilobectomy, pneumonectomy).
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2019-01-29 (Actual); Primary Completion 2021-03-01 (Actual); Study Completion 2021-08-01 (Actual)

PRIMARY OUTCOMES:
PAAL after pulmonary resection surgery | 5 days after operation
  End of bubbling is assessed by the nursing team in charge of the patient in accordance with the current practice (no bubbling at forced expiration), and validated by the physician in charge.

SECONDARY OUTCOMES:
clinical features | up to 28 days after the pulmonary resection surgery
  Collection of clinical features to identify risk factors for PAAL

CONTACTS AND LOCATIONS:
Overall Officials: Pierre SENTENAC, Dr, Principal Investigator — University Hospital, Montpellier
Locations (1):
- Department of Anesthesie Reanimation, Montpellier, France

IPD SHARING:
Plan to Share IPD: No